CLINICAL TRIAL: NCT02219282
Title: A Comparison of Laryngeal Mask UniqueTM in Denticulate and Edentulate Geriatric Patients
Brief Title: Geriatric Patients and Laryngeal Mask Unique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Anaesthesiology and Reanimation, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2010/08-15
Record Dates: First submitted 2014-07-31; First posted 2014-08-18 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Anaesthesia
Keywords: laryngeal mask airway, edentulate geriatric patients

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Dentulous (Active Comparator): Laryngeal Mask Unique insertion
  Interventions: Other: Laryngeal Mask Unique insertion
- Group Edentulous (Experimental): Laryngeal Mask Unique insertion
  Interventions: Other: Laryngeal Mask Unique insertion

INTERVENTIONS:
Other: Laryngeal Mask Unique insertion — Before insertion the laryngeal mask used in daily routine (Laryngeal Mask Unique) was lubricated with a water-based gel and the cuff was completely deflated. After induction when BIS values were between 40 and 60 and sufficient chin relaxation was obtained for patients weighing less than 50 kg no. 3 LMU, for those between 50-90 kg no. 4 and for patients above 90 kg no. 5 LMU was inserted by an anesthetist with more than three years experience.

SUMMARY:
As a result of rises in living standards quality of life is progressively increasing. Combined with developments in anesthesia, surgical techniques and medication allowing more difficult and complicated interventions to be carried out, elderly patients are encountered more often in daily anesthetic practice.Reduced tone in the upper airway of geriatric patients increases the possibility of airway obstruction. In old patients with no teeth, sunken cheeks may make ventilation with a mask ineffective; perhaps even impossible.

In addition to our observations that Laryngeal mask (LM) is more difficult to place in older patients, in the literature there are very few studies on the use of LM in older patients. Sixty percent of patients over the age of 65 have no teeth. Ventilation with a mask is more difficult for patients without teeth compared to those with teeth. Laryngeal mask is an alternative airway device for patients without teeth when the face mask does not sit correctly.

The aim of this study is primarily to measure the success of placement on first try, ease and duration of insertion and oropharyngeal leak pressure of laryngeal mask Unique (LMU) in patients 65 years of age and above dentulous and edentulous elderly patients. The secondary aim is to compare the effects on the hemodynamic response occurring during placement.

DETAILED DESCRIPTION:
This study received permission from Dokuz Eylül University Medical Faculty Ethics Committee and informed consent was obtained from the patients. Sixty-six patients above the age of 65 with American Society of Anesthesiologists (ASA) physiological classification group I-III, undergoing elective surgery and with indications for laryngeal mask placement participated in this prospective, and double bland study.

Patients taken to the operating room were monitored for heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), electrocardiography (ECG-Derivation II), and peripheral oxygen saturation (SpO2) before anesthesia induction. Depth of anesthesia was evaluated with a bispectral index monitor. The patients were preoxygenated with 6 L.min-1 oxygen through a face mask for 3 minutes. For anesthesia induction 0.02 mg.kg-1 midazolam, 1-2 μg.kg-1 fentanyl and 1-2 mg.kg-1 propofol were used. Afterwards patients were given mask ventilation with 100% oxygen. Before laryngeal masks were inserted they were prepared by being lubricated with water-based gel and the cuffs were completely deflated.

After induction agents were administered when BIS values were between 40-60 and sufficient chin relaxation was obtained LMU was inserted according to the standard methods determined by Brain. The LMU size was chosen based on the patient's body weight; those from 30-50 kg used no. 3, from 50-70 kg used no. 4 and those from 70-100 kg used no 5 LMU. During attempts depending on the patient reaction and to keep the BIS values 40-60, an additional dose of 0.5 mg/kg propofol was administered.

The cuffs of the laryngeal mask were inflated and held at 60 centimeters of water. After the operation before the LM was removed the cuff inner pressure was measured again and recorded. The success of the first attempt at insertion of the laryngeal mask was recorded. During placement in cases with 3 unsuccessful attempts, patients were intubated to provide airway management.

Anesthesia was maintained with a 50% O2/air mix with 1.5-2.5% sevoflurane. Concentration of sevoflurane was set to keep the bispectral index value below 40.

Systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP), heart rate (HR) and bispectral index values (BIS) were recorded before anesthesia induction, before LM insertion and in the 1st, 2nd, 3rd and 5th minutes after LM insertion was confirmed.

The time for successful insertion was defined as the duration from mouth opening to first successful ventilation and recorded. The number of insertion attempts and ease of insertion were recorded.

Criteria indicating successful laryngeal mask placement:

1. Waves with square shape on capnogram
2. Easy ventilation with respiration balloon and observed chest movement
3. No ventilation leak with approximately 20 centimeters of water positive pressure Evaluation of ease of insertion based on likert scala (1-4 point from easy to unsuccessful).

After laryngeal mask insertion, the oropharyngeal leak test was conducted by a researcher unaware of whether the patients had teeth or not. To complete the test after the expiring valve was shut fresh gas flow was reduced to 3 L.min-1. When the sound of a leak was heard from the mouth the airway pressure value (OLP) was recorded. During this test airway pressure was not allowed to rise above 40 centimeters of water. From the start of the operation to the end, the patients were monitored for hypoxia (SpO2 falling below 90%) and laryngospasm. In cases where the third attempt at LM insertion was unsuccessful, if the SpO2 values fell below 90% at any time in the study or if laryngospasm developed, the patients were excluded from the study.

The duration of use of laryngeal mask (duration from insertion to removal) in both groups were recorded. After the laryngeal mask was removed it was evaluated for traces of blood. When leaving the recovery unit and 24 hours later throat pain, dysphonia and dysphagia were evaluated. Throat pain was evaluated using the VAS-10 (visual analogue scale).

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 65
* ASA I-III
* Undergoing elective surgery

Exclusion Criteria:

* Patients with recent history of upper respiratory infection
* Obese patients with body-mass index above 35 kg/m2
* Symptomatic hiatus hernia
* Severe gastroesophageal reflux
* Those with low pulmonary compliance or high airway resistance (morbid obesity, lung disease)
* Throat pain, dysphagia and dysphonia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SEMİH KUCUKGUCLU, M.D., Study Director — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation, Izmi̇r, Narlıdere, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Dentulous | Group Edentulous
Started | 33 | 33
Completed | 32 | 32
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Dentulous | Group Edentulous | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 33 | 33 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  Turkey | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Laryngeal Mask Placement
Description: The aim of this study is primarily to measure the success of placement on first try in dentulous and edentulous elderly patients for success of placement on first try.
Time Frame: Baseline
Population: For one patient in each group, dentulous and edentulous, insertion of the LMU was unsuccessful on the third attempt, and these patients were intubated; therefore, these two patients were excluded from the study and were not included in the statistical analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group Dentulous | Group Edentulous
Number analyzed (Participants) | 32 | 32
Participants
  First Attempt | 26 | 20
  Second Attempt | 6 | 11
  Third attempt | 0 | 1

2. Secondary Outcome: Oropharyngeal Leak Pressure
Description: Oropharyngeal leak pressure (cm H20) in dentulous and edentulous elderly patients.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm H20
Arm/Group | Group Dentulous | Group Edentulous
Number analyzed (Participants) | 32 | 32
cm H20 | 21.75 (4.62) | 20.75 (5.04)

3. Secondary Outcome: Haemodynamic Response to Insertion of Airway Device.
Description: Mean blood pressure (MBP) (mmHg) were recorded in both groups.
Time Frame: Before anesthesia induction, before laryngeal mask insertion and in the 1st, 2nd, 3rd and 5th minutes after laryngeal mask insertion
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group Dentulous | Group Edentulous
Number analyzed (Participants) | 32 | 32
mmHg
  Before anesthesia induction | 94.3 (10) | 95.1 (12)
  before laryngeal mask insertion | 80.1 (8) | 80.2 (9)
  1 minutes after laryngeal mask insertion | 80.1 (5) | 79.2 (6)
  2 minutes after laryngeal mask insertion | 70.2 (8) | 73.1 (6)
  3 minutes after laryngeal mask insertion | 71.2 (7) | 70.3 (8)
  5 minutes after laryngeal mask insertion | 70.4 (7) | 72.6 (8)

4. Secondary Outcome: Ease of Placement Laryngeal Mask
Description: Ease (according to Likert scale 1-4 point from easy to diffucult).
Time Frame: During Laryngeal mask placement
Measure: Count of Participants; unit: Participants
Groups:
- Dentulous; Edentuolus: Laryngeal Mask Unique insertion
  Laryngeal Mask Unique insertion: Before insertion the laryngeal mask used in daily routine (Laryngeal Mask Unique) was lubricated with a water-based gel and the cuff was completely deflated. After induction when BIS values were between 40 and 60 and sufficient chin relaxation was obtained for patients weighing less than 50 kg no. 3 LMU, for those between 50-90 kg no. 4 and for patients above 90 kg no. 5 LMU was inserted by an anesthetist with more than three years experience
Arm/Group | Dentulous | Edentuolus
Number analyzed (Participants) | 32 | 32
Participants
  1 | 30 | 25
  2 | 2 | 7

5. Secondary Outcome: Insertion Time of Laryngeal Mask
Description: Duration of insertion (second) Laryngeal Mask;second
Time Frame: During placement of Laryngeal Mask
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Dentilous Group; Edentulous Group: Laryngeal Mask Unique insertion
  Laryngeal Mask Unique insertion: Before insertion the laryngeal mask used in daily routine (Laryngeal Mask Unique) was lubricated with a water-based gel and the cuff was completely deflated. After induction when BIS values were between 40 and 60 and sufficient chin relaxation was obtained for patients weighing less than 50 kg no. 3 LMU, for those between 50-90 kg no. 4 and for patients above 90 kg no. 5 LMU was inserted by an anesthetist with more than three years experience
Arm/Group | Dentilous Group | Edentulous Group
Number analyzed (Participants) | 32 | 32
seconds | 14.40 (4.80) | 13.43 (4.11)

ADVERSE EVENTS:
Arm/Group | Group Dentulous | Group Edentulous
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No